CLINICAL TRIAL: NCT00560183
Title: A Placebo-controlled, Randomized, Double-blind Study of the Safety and Efficacy of Q8003 in the Management of Post-bunionectomy Pain
Brief Title: Efficacy and Safety of Q8003 in the Management of Post-bunionectomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q8003-007
Record Dates: First submitted 2007-11-14; First posted 2007-11-19 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: Acute; Bunionectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — MoxDuo; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Q8003 (morphine sulfate and oxycodone hydrochloride)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q8003 (morphine sulfate and oxycodone hydrochloride) — Capsules, four different mg dosage strengths
  Arms: 1
Drug: Placebo — Capsules
  Arms: 2

SUMMARY:
This study will explore the efficacy and safety of a fixed dose combination of morphine and oxycodone for management of acute postoperative pain. The study will explore the efficacy dose response and dosing interval required to maintain adequate analgesia at each tested dosage strength.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, rising-dose/by-cohort study of the efficacy and safety of Q8003 in inpatients with acute pain following unilateral bunionectomy surgery. Patients in each dosing group will receive either Q8003 (approximately 50 per dosing group) or placebo (approximately 13 per dosing group), determined by random sequential assignment and blinded to patients and managing Investigators. Dosing groups will be enrolled sequentially in ascending order; only one dosing group will be open at a time for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for bunionectomy surgery and is willing to stay in the study center for at least 48 hours from the initial dose of study medication post surgery.
* Females must be non-pregnant, non-lactating, and practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥12 months).
* Patient has normal laboratory values or abnormal values judged not clinically significant by the Investigator for clinical chemistry and hematology (< 1.5 ULN).
* Patient is in general good health based on physical examination, medical history and clinically acceptable results for the following assessments: vital signs and a 12-lead electrocardiogram (ECG).
* Patient gives written informed consent and is able to understand the requirements of the study, adhere to the study restrictions, and be available for the required follow-up assessment.

Exclusion Criteria:

* Patient has a current acute or chronic disease that would interfere with evaluations of postoperative Q8003 efficacy or safety.
* Patient has a history of poor tolerance to short term opiate use in prior surgeries, based on patient self-report.
* Patient used opiates continuously (including tramadol) for more than five days in the past year.
* Patient has a history of pulmonary, cardiovascular, neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that, in the opinion of the Investigator, would jeopardize the patient's well-being by participation in this study.
* Patient has positive HIV serology or signs of HIV infection or AIDS.
* Patient has positive HBsAg or HCV antibody.
* Patient is currently receiving any medications that are not at a stable dose (the same dose for >2 month prior to date of surgery).
* Patient is currently receiving muscle relaxants, antipsychotic drugs, monoamine oxidase inhibitors, or any medications for the treatment of depression.
* Patient has used systemic corticosteroids within previous fourteen (14) days.
* Patient was dosed with another investigational drug within 30 days prior to the Screening Visit.
* Patient has current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).
* Patient has a history of abusing licit or illicit drug substances within five (5) years of study entry.
* Patient is obese with a body mass index >32.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity scores from baseline | 48 hours

SECONDARY OUTCOMES:
Appropriate dosing interval for each tested dose level | 48 hours
Safety: incidence of opioid-related adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Warren Stern, Ph.D., Study Director — QRxPharma Inc.
Locations (6):
- United States (6):
  - Advanced Clinical Research Institute, Anaheim, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Advanced Regional Center for Foot and Ankle Care, Altoona, Pennsylvania
  - Scirex Research Center, Houston, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah